CLINICAL TRIAL: NCT06286774
Title: Sleep as a Mechanism of Change in Alcohol Use Outcomes Among Heavy-Drinking Adults
Brief Title: Sleep as a Mechanism of Change in Alcohol Use
Acronym: ReTRAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Mary E Miller, Associate Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2096884
Record Dates: First submitted 2024-02-02; First posted 2024-02-29 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Insomnia; Alcohol; Harmful Use
Keywords: alcohol; drinking; sleep; insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to Cognitive Behavioral Therapy for Insomnia (CBT-I) or waitlist control.
Who Masked: Investigator, Outcomes Assessor
Masking Description: PI Miller and study therapists will be blinded to assessment outcomes, and assessment RAs will be blinded to participant condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-I (Experimental): Individual Cognitive Behavioral Therapy for Insomnia (CBT-I) delivered once a week for five (5) weeks.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- Waitlist control (No Intervention): Control participants will receive CBT-I at the end of the study.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — Cognitive Behavioral Therapy for Insomnia (CBT-I). Participants assigned to the CBT-I condition will attend 1-hour individual sessions of CBT-I once a week for five weeks. Consistent with clinical guidelines (Schutte-Rodin, Broch, Buysse, Dorsey, & Sateia, 2008), treatment will include stimulus control (e.g., limit use of bed to sleep or sexual activity, get out of bed if lying awake for more than 20 minutes), sleep restriction (limit time in bed to amount of time spent sleeping on a typical night), sleep hygiene (e.g., avoid exercise within 2 hours of bedtime, create cool and dark sleep environment), relaxation training, and cognitive restructuring.
  Other Names: CBT-I
  Arms: CBT-I

SUMMARY:
This project aims to evaluate improvement of insomnia as a mechanism of improvement in alcohol use outcomes.

DETAILED DESCRIPTION:
Heavy alcohol use is prevalent in the United States and results in significant physical and psychological burden. One in 10 adults in the United States reports binge drinking on a weekly basis, and few are willing to seek mental health treatment. Thus, additional strategies are needed to engage and treat individuals at risk for alcohol-related harm. Half of those who screen positive for hazardous drinking report clinically significant symptoms of insomnia. Insomnia tends to be less stigmatized than other mental health disorders, and it is one condition for which the field has highly efficacious treatment. Thus, one potential strategy to engage individuals in mental health treatment and reduce the burden of alcohol use in the United States is to target insomnia. This project aims (1) to examine change in insomnia as a mediator of insomnia treatment effects on alcohol use outcomes and sex as a moderator of those effects and (2) to identify mechanisms linking change in insomnia to alcohol use outcomes. Adults who drink alcohol and have insomnia will be randomly assigned to Cognitive Behavioral Therapy for Insomnia (CBT-I, n=112) or waitlist control (WLC, n=112). Outcomes will be assessed weekly during treatment, at the end of the active intervention period (post-treatment), and at 1-, 3-, and 6-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* report heavy drinking in a typical week in the past month
* meet DSM-5 criteria for Alcohol Use Disorder
* meet DSM-5 and research diagnostic criteria for Insomnia Disorder

Exclusion Criteria:

* ≥50 years
* unable to provide informed consent
* report contraindications for CBT-I (mania or seizure disorder)
* moderate to severe sleep apnea that is untreated
* have symptoms requiring immediate clinical attention (e.g., psychosis, suicide plan)
* are already receiving behavioral treatment for insomnia or alcohol use

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 256 (Estimated)
Dates: Start 2024-03-02 (Actual); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Insomnia Symptoms | Change from baseline to mid-treatment (week 4) to post-treatment (week 6) to 1-, 3-, and 6-month follow-ups
  Assessed using Insomnia Severity Index (ISI). Response options range from 0 (not at all worried) to 4 (very much worried), with total scores ranging from 0 to 28 and higher scores indicating more severe insomnia.
Drinking quantity | Change from baseline to post-treatment (week 6) to 1-, 3-, and 6-month follow-ups
  Assessed using Timeline Followback and Daily Drinking Questionnaire. Typical weekly drinking quantity estimates will be summed to create a "drinks per week" total score, which will be used as our outcome variable.
Alcohol-related consequences | Change from baseline to post-treatment (week 6) to 1-, 3-, and 6-month follow-ups
  Assessed using the Drinker Inventory of Consequences (DrINC). Scores range from 0 to 120, with higher scores indicating more consequences. The common consequence subscale scores range from 0 to 18.

SECONDARY OUTCOMES:
Treatment willingness (alcohol) | Change from baseline to post-treatment (week 6)
  Assessed using a modified Treatment Willingness Scale. Participants rate their agreement with the statement that they would seek treatment for 5 medical and 5 mental health conditions if they experienced problems related to them. Willingness to seek alcohol or drug treatment is assessed on a 0-5 scale, with higher scores indicating greater willingness.
Alcohol craving | Change from baseline to post-treatment (week 6) to 1-, 3-, and 6-month follow-ups
  Assessed using the Penn Alcohol Craving Scale (PACS). PACS evaluates thoughts about drinking by assessing the duration, frequency, and intensity of such thoughts. Scores range 0-30, with higher scores indicating more severe craving.
Negative emotionality | Change from baseline to post-treatment (week 6) to 1-, 3-, and 6-month follow-ups
  Negative emotionality will be assessed as a latent construct of mood, anxiety, depression, PTSD symptoms, and difficulties with emotion regulation. Changes in individual symptoms will be reported for descriptive purposes.
Response inhibition | Change from baseline to post (week 6) to 3-month follow-up
  Assessed using the Stroop Task. Average reaction time (RT; measured from color word/color rectangle stimuli onset until a response is made) on correct trials for each trial type (control trials, congruent trials, incongruent trials) were computed as the outcomes of interest. Higher RTs indicate worse performance.
Working memory | Change from baseline to post (week 6) to 3-month follow-up
  Assessed using the N-Back Task. The dependent measure is the proportion of correct responses (yes and no) across all four blocks. Omissions are counted as errors.
Delay discounting | Change from baseline to post-treatment (week 6) to 1-, 3-, and 6-month follow-ups
  Assessed using the Monetary Choice Questionnaire (MCQ). Participants indicate if they would rather receive a smaller amount of money now or a greater amount of money in a specified amount of time (e.g., 100 days, 2 days). The MCQ is scored using a logarithmic subject-specific discount rate (k variable). Higher k values indicate a greater preference for smaller, immediate rewards over larger, delayed reward.
Alcohol to help with sleep | Change from baseline to post-treatment (week 6) to 1-, 3-, and 6-month follow-ups
  Assessed using daily sleep diaries. The outcome will be percentage of days using alcohol to help with sleep.
Heartrate variability | Change from baseline to post-treatment (week 6) to 1-, 3-, and 6-month follow-ups
  Assessed using Fitbit Charge 6. Heart-rate variability (HRV) is an indicator of activity in the autonomic nervous system that quantifies changes in intervals between heart beats. In general, HRV increases with increasing parasympathetic activity, then plateaus and decreases with increasing sympathetic activity.
Dysfunctional Beliefs and Attitudes about Sleep Scale | Change from baseline to post-treatment (week 6) to 1-, 3-, and 6-month follow-ups
  Assessed using the revised Dysfunctional Beliefs and Attitudes about Sleep Scale. Responses range from 0 to 70, with higher scores indicating more dysfunctional beliefs.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States